CLINICAL TRIAL: NCT07320638
Title: Expression of Trim25 in Peripheral Blood Mononuclear Cells of Patients With Sepsis and Non-sepsis and Its Relationship With the Prognosis of Patients With Sepsis
Brief Title: TRIM25 in Septic Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sepsis-2021-278; 81900073 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Genes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-sepsis patients: Sepsis patients
  Interventions: Diagnostic Test: Gene and Inflammatory Marker Analysis in Sepsis

INTERVENTIONS:
Diagnostic Test: Gene and Inflammatory Marker Analysis in Sepsis — 1.Sepsis Group:
  1. SOFA score >=2;
  2. Aged 18-70 years male and female;
  3. Hospitalization. 2.Non-sepsis Group:
  (1) Healthy adults; (2) Aged 18-70 years male and female.

SUMMARY:
Sepsis is a life-threatening condition caused by the body's overwhelming response to infection, which can lead to organ damage and failure. The goal of this observational study is to better understand the underlying biological changes that occur in patients with sepsis compared to those who do not have the condition.

We will collect peripheral blood samples from patients diagnosed with sepsis and from non-sepsis control participants. From these samples, we will isolate peripheral blood mononuclear cells (PBMCs) and serum.

We will then analyze these components to measure the activity of specific genes and the levels of key inflammatory factors (cytokines).

The information we gather will help researchers identify molecular and inflammatory markers associated with sepsis. This knowledge is crucial for developing new and more effective methods for diagnosing and treating this critical illness.

ELIGIBILITY:
Inclusion Criteria:

* 1. SOFA score >=2; 2. Aged 18-70 years male and female; 3. Hospitalization.

Exclusion Criteria:

* 1. Immune system disease, such as HIV; 2. Disease that possibly affect the function of immune system, such as tumor and chronic viral infection; 3. Patients that treated with massive cortical hormone (>200mg/d) or immunosuppressant; 4. Pregnant or lactation women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of two primary, non-overlapping groups of adult participants recruited from the hospital setting:
  Sepsis Patient Cohort (Case Group): Adult patients (aged 18 years or older) who are diagnosed with Sepsis based on the Sepsis-3 clinical criteria (or the most current widely accepted clinical definitions) upon admission to the Intensive Care Unit (ICU) or general ward.
  Non-Sepsis Control Cohort (Control Group): Adult patients (aged 18 years or older) who are admitted to the hospital with non-infectious conditions or healthy volunteers, provided they do not meet the criteria for sepsis or severe infection at the time of enrollment.
  The enrollment process for both groups will be observational, involving the collection of a single peripheral blood sample for the isolation of peripheral blood mononuclear cells (PBMCs) and serum, as well as collection of relevant clinical data.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
TRIM25 in PBMCs | From 2021.12 to 2026.06
  We will collect peripheral blood mononuclear cells (PBMCs) from both sepsis patients and non-sepsis control patients to compare the expression level of the TRIM25 gene in these cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai JiaoTong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided